CLINICAL TRIAL: NCT00110149
Title: A Phase II Study of Yttrium-90-Labeled Ibritumomab Tiuxetan (Zevalin) Radioimmunotherapy as First Line Treatment in Indolent Non-Hodgkin's Lymphoma
Brief Title: Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company withdrew drug supply
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Robin Joyce, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004P000044; CDR0000409723 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02445 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; stage I grade 1 follicular lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; splenic marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan (Experimental): Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
  Interventions: Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others, such as yttrium Y 90 ibritumomab tiuxetan, find cancer cells and help kill them or carry cancer-killing substances to them without harming normal cells. Giving rituximab together with yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with yttrium Y 90 ibritumomab tiuxetan works in treating patients with indolent non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine 12-week overall and complete response rate in patients with indolent non-Hodgkin's lymphoma treated with rituximab and yttrium Y 90 ibritumomab tiuxetan as first-line treatment.

Secondary

* Determine 1-year event-free survival of patients treated with this regimen.
* Determine time to progression and time to next antilymphoma therapy in patients treated with this regimen.
* Determine the molecular response rate in patients treated with this regimen.
* Determine the hematological and non-hematological toxicity of this regimen in these patients.
* Assess the quality of life of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive rituximab IV followed, no more than 4 hours later, by indium In 111 ibritumomab tiuxetan (for imaging) IV over 10 minutes on day 1. If biodistribution is acceptable, patients receive rituximab IV followed, no more than 4 hours later, by a single dose of yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 7, 8, or 9 in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, weeks 6, 10, and 14, every 3 months for 2 years, and then every 6 months for 2 years.

After completion of study treatment, patients are followed weekly for 3 months, every 3 months for 2 years, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 18-28 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed indolent non-Hodgkin's lymphoma (NHL), including 1 of the following histologic subtypes:

  * Grade1 or 2 follicular lymphoma
  * Small lymphocytic lymphoma (SLL)
  * Marginal zone B-cell lymphoma
* CD20-positive disease confirmed by immunohistochemistry or flow cytometry
* Bidimensionally measurable disease

  * At least 1 lesion measuring ≥ 2.0 cm in a single dimension by CT scan
* Less than 25% bone marrow involvement with lymphoma by bilateral iliac crest bone marrow aspiration and biopsy within the past 6 weeks
* No clinically significant impaired bone marrow reserve as evidenced by any of the following:

  * Hypocellular marrow, as evidenced by 1 of the following:

    * ≤ 15% cellularity
    * Marked reduction in bone marrow precursors
  * Platelet count < 100,000/mm^3
  * Absolute neutrophil count < 1,500/mm^3
  * History of failed stem cell collection
  * Prior myeloablative therapy
* No greater than 5,000/mm^3 circulating tumor cells in peripheral blood
* Requires antilymphoma therapy, as indicated by any of the following:

  * Systemic symptoms
  * B symptoms
  * Cytopenias
  * Malaise
  * Organ compromise
  * Discomfort
  * Pain
  * Disfigurement
  * Rapidly progressive disease
  * Undue anxiety related to not receiving treatment
* No transformation to intermediate or high-grade NHL
* No known brain metastases or CNS involvement by lymphoma NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2 OR
* WHO 0-2 OR
* Karnofsky 70-100%

Life expectancy

* More than 3 months

Hematopoietic

* See Disease Characteristics
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Lymphocyte count < 5,000/mm^3 (for patients with SLL )

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal

Renal

* Creatinine ≤ 2.0 mg/dL OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Immunologic

* No anti-murine antibody reactivity (in patients with prior exposure to murine antibodies or proteins)
* No ongoing or active infection
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to yttrium Y 90 ibritumomab tiuxetan

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 1 year after study treatment
* No other active malignancy except non-melanoma skin cancer
* No other serious nonmalignant disease that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior pegfilgrastim
* More than 2 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior external beam radiotherapy to > 25% of active bone marrow (involved field or regional)

Surgery

* More than 4 weeks since prior major surgery except diagnostic surgery

Other

* No prior systemic antilymphoma therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No other concurrent antilymphoma therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-05; Primary Completion 2012-05 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Joyce, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 patients were recruited and signed consent. 3 patient were ineligible and were not treated. The total number treated is nine
Period: Overall Study
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Started | 12 (total number that signed consent to be screened.)
Received Treatment | 9 (total number of patient that passed screening and received treatment.)
Completed | 9
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response, Unconfirmed Complete Response, and Partial Response) at 12 Weeks
Description: INTERNATIONAL WORKSHOP RESPONSE CRITERIA FOR NON HODGKIN'S LYMPHOMA
  Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, et al. Report of an international workshop to standardize response criteria for non Hodgkin's lymphoma. J Clin Oncol 1999;17(4):1244-53.
Time Frame: 14 weeks
Population: The trial closed prematurely secondary to the company that produced the agent being sold to another company and the agent not being available to treat the full number of patients in this trial.
Measure: Count of Participants; unit: Participants
Groups:
- Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan: patient un treated NHL, who were then treated with the Rituximab and Y-90 Ibritumomab Tiuxetan.
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 9
Participants
  CR | 9
  PR | 0
  PD | 0
Statistical Analysis 1: Comparison: Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan; Test type: Other — As the study was not able to be completed the simple number of patients per outcome is listed; The trial was to measure the response rate and EFS of patients but the manufacturer of the investigational agent closed and sold the agent to a new company so the trial was not able to be completed

2. Primary Outcome: EFS
Description: Event = Death, second malignancy , disease progression.
Time Frame: 1 year
Population: The study was terminated early
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 9
Participants
  Progression | 3
  alive in remission | 5
  Second malignancy | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan (N=9)
neutropenia (Blood and lymphatic system disorders) | 4 (4) — grade 3 neutropenia

LIMITATIONS AND CAVEATS:
This trial was stopped abruptly when the makers of the investigational agent sold the company and the agent was not available for a significant period of time. Attempts were made to follow all patients for 12 months after treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No